CLINICAL TRIAL: NCT04264819
Title: A One-year, Single-arm, Open-label, Multicenter Study Assessing the Effect of Brolucizumab on Disease Control in Adult Patients With Suboptimal Anatomically Controlled Neovascular Age-related Macular Degeneration (SWIFT)
Brief Title: Study of Brolucizumab in Adult Patients With Suboptimal Anatomically Controlled Neovascular Age-related Macular Degeneration
Acronym: SWIFT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRTH258AFR03; 2019-004145-33 (EudraCT Number)
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Results first posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-09

CONDITIONS: Neovascular Age-Related Macular Degeneration
Keywords: Macular degeneration; age-related macular degeneration (ARMD); vision loss; macula damage; retina damage; dry macular degeneration; wet macular degeneration; AMD; diabetic macular edema; DME; neovascular age-related macular degeneration; nAMD; retinal vein occlusion; RVO; wetAMD; neovascular; choroidal neovascularization; disease control
MeSH Terms: conditions — Macular Degeneration; Vision Disorders; Geographic Atrophy; Wet Macular Degeneration; Retinal Vein Occlusion; Choroidal Neovascularization | interventions — brolucizumab

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RTH258/Brolucizumab (Experimental): This is a single arm study in which all patients will be treated with brolucizumab 6mg; 3 loading injections (at Screening/Baseline, week 4 and week 8) followed by treat-to-control phase with adjustable treatment frequency based on disease activity from every 8 to up to 16 weeks; last treatment at week 44/46 based on the treatment regimen.
  Interventions: Drug: RTH258/Brolucizumab

INTERVENTIONS:
Drug: RTH258/Brolucizumab — Brolucizumab is a new generation of anti-VEGF (vascular endothelial growth factor). All patients will be treated with brolucizumab 6mg: 3 loading injections (at Screening/Baseline, Week 4 and Week 8), followed by Treat-to-Control regimen up to Week 44/46.

SUMMARY:
Neovascular age-related macular degeneration is characterized by the presence of choroidal neovascularization (CNV), which consists of abnormal blood vessels originating from the choroid that can lead to hemorrhage, fluid exudation, and fibrosis, resulting in photoreceptor damage and vision loss.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label, multicenter study to evaluate the efficacy and safety of brolucizumab 6 mg in pretreated suboptimal anatomically controlled patients with neovascular age-related macular degeneration (nAMD).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must provide written informed consent before any study-related procedures are performed.
2. Patients must be 50 years of age or older at Screening/Baseline.

   Study eye:
3. Active CNV lesions secondary to nAMD diagnosed < 18 months prior to Screening/Baseline that affect the central subfield, including retinal angiomatous proliferation (RAP) with a CNV component, confirmed by presence of active leakage from CNV seen by FA and sequelae of CNV, e.g. pigment epithelial detachment (PED), subretinal hemorrhage or sub RPE hemorrhage, blocked fluorescence, or macular edema.
4. Previous treatment with only one licensed anti-VEGF drug (i.e. Lucentis®, Eylea®) with a ≥ Q4 and ≤ Q8 treatment (treatment interval of 26 to 62 days inclusive) with licensed anti-VEGF (a minimal washout period of at least 4 weeks / 26 days is required). Patients must have received at least 3 injections of this anti-VEGF in the 6 months prior to Screening/Baseline.
5. Presence of residual fluid (IRF or SRF that affects the central subfield under, as seen by OCT)
6. BCVA score must be ≤ 83 and ≥ 38 letters at an initial testing distance of 4 meters starting distance using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity charts at Screening/Baseline.

Exclusion Criteria:

Ocular conditions

1. Any active intraocular or periocular infection or active intraocular inflammation (e.g. infectious conjunctivitis, keratitis, scleritis, endophthalmitis, infectious blepharitis), in either eye at Screening/Baseline.
2. Presence of amblyopia, amaurosis, or ocular disorders in the fellow eye with BCVA < 35 ETDRS letters at Screening/Baseline (except when due to conditions whose surgery may improve visual acuity, e.g. cataract).
3. Medical history of intraocular inflammation and/or retinal vascular occlusion within 12 months prior to Screening/Baseline

   Study eye
4. Poor quality of OCT image at Screening/Baseline.
5. Atrophy or fibrosis involving the center of the fovea in the study eye, as assessed by CFP and fundus autofluorescence (FAF).
6. The total area of fibrosis or subretinal blood affecting the foveal center point comprising ≥ 50% of the lesion area in the study eye.
7. Concomitant conditions or ocular disorders in the study eye, including retinal diseases other than nAMD, that, in the judgment of the Investigator, could require medical or surgical intervention during the course of the study to prevent or treat visual loss that might result from that condition, or that limits the potential to gain visual acuity upon treatment with the investigational product.
8. Structural damage within 0.5 disc diameter of the center of the macula in the study eye, e.g. vitreomacular traction, epiretinal membrane, RPE rip/tear scar, laser burn, at the time of Screening/Baseline that in the Investigator's opinion could preclude visual function improvement with treatment.
9. Current vitreous hemorrhage or history of vitreous hemorrhage in the study eye within 4 weeks prior to Screening/Baseline.
10. Uncontrolled glaucoma in the study eye defined as IOP > 25 mmHg on medication or according to the Investigator's judgment, at Screening/Baseline.
11. Aphakia and/or absence of the posterior capsule in the study eye. Ocular treatments (study eye)
12. Patient has received any investigational treatment for nAMD (other than vitamin supplements) in the study eye at any time.
13. Previous use of intraocular or periocular of corticosteroids in the study eye within the 6 month period prior to Screening/Baseline.
14. Previous penetrating keratoplasty or vitrectomy at any time prior to Screening/Baseline.
15. History or evidence of the following in the study eye within the 90-day period prior to Screening/Baseline:

    * Intraocular or refractive surgery.
    * Previous panretinal and peripheral laser photocoagulation.
    * Previous macular surgery or other intraocular surgical intervention
16. Previous laser treatment for nAMD including photodynamic therapy (PDT) laser at any time prior to Screening/Baseline.
17. Previous treatment with investigational drugs.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2023-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (40):
- France (40):
  - Novartis Investigative Site, Nice, Cedex1
  - Novartis Investigative Site, Rennes, FRA
  - Novartis Investigative Site, Saint-Cyr-sur-Loire, Indre Et Loire
  - Novartis Investigative Site, Lyon, Rhone
  - Novartis Investigative Site, Bobigny, Seine Saint Denis
  - Novartis Investigative Site, Aix-en-Provence
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Colmar
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, La Rochelle
  - Novartis Investigative Site, La Valette-du-Var
  - Novartis Investigative Site, Le Chesnay
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Melun
  - Novartis Investigative Site, Montargis
  - Novartis Investigative Site, Montauban
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Mulhouse
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Perpignan
  - Novartis Investigative Site, Plérin
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Rueil-Malmaison
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Saint-Jean
  - Novartis Investigative Site, Saint-Jean-de-Védas
  - Novartis Investigative Site, Saint-Martin-des-Champs
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tours
  - Novartis Investigative Site, Vincennes

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Bodaghi B, Souied EH, Tadayoni R, Weber M, Ponthieux A, Kodjikian L. Detection and Management of Intraocular Inflammation after Brolucizumab Treatment for Neovascular Age-Related Macular Degeneration. Ophthalmol Retina. 2023 Oct;7(10):879-891. doi: 10.1016/j.oret.2023.06.009. Epub 2023 Jun 19. PMID 37343623

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Before inclusion, patients underwent a 4-to-8-Week Washout Period (from 26 to 62 days) from the last administration of a licensed anti-VEGF drug (i.e., Lucentis®, Eylea®).
Groups:
- RTH258/Brolucizumab: This is a single arm study in which all patients are treated with brolucizumab 6mg; 3 loading injections (at Screening/Baseline, week 4 and week 8) followed by treat-to-control phase with adjustable treatment frequency based on disease activity from every 8 to up to 16 weeks; last treatment at week 44/46 based on the treatment regimen.
Period: Overall Study
Arm/Group | RTH258/Brolucizumab
Started | 295
Full Analysis Set (FAS) | 289 (The FAS comprised all patients who received at least one intravitreal (IVT) injection of study treatment and did not have any protocol deviations with impact.)
Completed | 249
Not Completed | 46
Not completed — Physician Decision | 19
Not completed — Adverse Event | 12
Not completed — Withdrawal by Subject | 11
Not completed — Lost to Follow-up | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 295
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 273
Age, Continuous [Mean (Standard Deviation); unit: Years] | 76.2 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183
  Male | 112
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With no Disease Activity at Week 16 in the Study Eye
Description: Disease activity criteria were assessed by the Investigator based on whether neovascular age-related macular degeneration (nAMD) was still active or had been re-activated. The disease was defined as active if at least one of the following criteria was observed:
  * Best-corrected visual acuity (BCVA) decrease ≥ 5 letters from the best value since Baseline due to disease activity
  * Any significant increase in central retinal thickness (CRT)
  * Retinal hemorrhage
  * Intraretinal fluid or sub-retinal fluid (SRF) due to disease activity (degenerative cysts allowed)
  * Increase of sub-retinal pigmented epithelium (RPE) fluid These criteria were for guidance only, Investigators could define disease activity based on their own assessment.
Time Frame: Week 16
Population: Full Analysis Set - The full analysis set (FAS) comprises all patients who received at least one IVT injection of study treatment without protocol deviation with impact and with an assessment of disease activity at Week 16.
Measure: Count of Participants; unit: Participants
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 217
Participants | 89

2. Secondary Outcome: Number of Patients With no Disease Activity at Week 48 in the Study Eye
Description: as for outcome 1
Time Frame: Week 48
Population: Full Analysis Set - The full analysis set (FAS) comprises all patients who received at least one IVT injection of study treatment without protocol deviation with impact and with an assessment of disease activity at Week 48.
Measure: Count of Participants; unit: Participants
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 196
Participants | 102

3. Secondary Outcome: Change From Baseline in CFST (Central Sub-Field Retinal Thickness) as Assessed by OCT (Optical Coherence Tomography) Over Time up to Week 48 in the Study Eye
Description: Central Subfield Thickness Assessed by Spectral domain optical coherence tomography (SD-OCT) from the central reading center.
Time Frame: Baseline, Weeks 4,8,16, 48
Population: Full Analysis Set - The full analysis set (FAS) comprises all patients who received at least one IVT injection of study treatment without protocol deviation with impact and had at least one valid post-baseline assessment.
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 258
μm
  Week 4 | -79.19 (79.874)
  Week 8 (n=227): number analyzed (Participants) | 227
  Week 8 (n=227) | -88.08 (91.505)
  Week 16 (n=220): number analyzed (Participants) | 220
  Week 16 (n=220) | -48.87 (84.345)
  Week 48 (n = 195): number analyzed (Participants) | 195
  Week 48 (n = 195) | -66.75 (101.496)

4. Secondary Outcome: Absence of IRF (Intraretinal Fluid), SRF (Subretinal Fluid), and Sub-RPE (Retinal Pigmented Epithelium) Fluid as Assessed by OCT Over Time up to Week 48 in the Study Eye
Description: Assessed by Spectral domain optical coherence tomography (SD-OCT) from the central reading center.
  At week 8, for 1 patient, the fluid assessment was performed, but result is unknown; at week 16, for 1 patient, the fluid assessment was performed, but result is unknown; at week 48, for 2 patients, the fluid assessment was performed, but result is unknown.
Time Frame: Baseline, Week 4, 8, 16, 48
Population: Full Analysis Set - The full analysis set (FAS) comprises all patients who received at least one IVT injection of study treatment without protocol deviation with impact
Measure: Count of Participants; unit: Participants
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 289
Participants
  Baseline - Intraretinal fluid | 104
  Baseline - Subretinal fluid | 245
  Baseline - Sub-RPE fluid | 204
  Baseline - Without any fluid (IRF/SRF) | 4
  Baseline - With any fluid (IRF/SRF) | 285
  Week 4 - Intraretinal fluid (n=260): number analyzed (Participants) | 260
  Week 4 - Intraretinal fluid (n=260) | 61
  Week 4 - Subretinal fluid (n=260): number analyzed (Participants) | 260
  Week 4 - Subretinal fluid (n=260) | 102
  Week 4 - Sub-RPE fluid (n=260): number analyzed (Participants) | 260
  Week 4 - Sub-RPE fluid (n=260) | 102
  Week 4 - Without any fluid (IRF/SRF) (n=260): number analyzed (Participants) | 260
  Week 4 - Without any fluid (IRF/SRF) (n=260) | 114
  Week 4 - With any fluid (IRF/SRF) (n=260): number analyzed (Participants) | 260
  Week 4 - With any fluid (IRF/SRF) (n=260) | 146
  Week 8 - Intraretinal fluid (n=229): number analyzed (Participants) | 229
  Week 8 - Intraretinal fluid (n=229) | 50
  Week 8 - Subretinal fluid (n=229): number analyzed (Participants) | 229
  Week 8 - Subretinal fluid (n=229) | 72
  Week 8 - Sub-RPE fluid (n=229): number analyzed (Participants) | 229
  Week 8 - Sub-RPE fluid (n=229) | 74
  Week 8 - Without any fluid (IRF/SRF) (n=229): number analyzed (Participants) | 229
  Week 8 - Without any fluid (IRF/SRF) (n=229) | 122
  Week 8 - With any fluid (IRF/SRF) (n=229): number analyzed (Participants) | 229
  Week 8 - With any fluid (IRF/SRF) (n=229) | 106
  Week 16 - Intraretinal fluid (n=222): number analyzed (Participants) | 222
  Week 16 - Intraretinal fluid (n=222) | 70
  Week 16 - Subretinal fluid (n=222): number analyzed (Participants) | 222
  Week 16 - Subretinal fluid (n=222) | 117
  Week 16 - Sub-RPE fluid (n=222): number analyzed (Participants) | 222
  Week 16 - Sub-RPE fluid (n=222) | 99
  Week 16 - Without any fluid (IRF/SRF) (n=222): number analyzed (Participants) | 222
  Week 16 - Without any fluid (IRF/SRF) (n=222) | 69
  Week 16 - With any fluid (IRF/SRF) (n=222): number analyzed (Participants) | 222
  Week 16 - With any fluid (IRF/SRF) (n=222) | 152
  Week 48 - Intraretinal fluid (n=198): number analyzed (Participants) | 198
  Week 48 - Intraretinal fluid (n=198) | 64
  Week 48 - Subretinal fluid (n=198): number analyzed (Participants) | 198
  Week 48 - Subretinal fluid (n=198) | 84
  Week 48 - Sub-RPE fluid (n=198): number analyzed (Participants) | 198
  Week 48 - Sub-RPE fluid (n=198) | 85
  Week 48 - Without any fluid (IRF/SRF) (n=198): number analyzed (Participants) | 198
  Week 48 - Without any fluid (IRF/SRF) (n=198) | 80
  Week 48 - With any fluid (IRF/SRF) (n=198): number analyzed (Participants) | 198
  Week 48 - With any fluid (IRF/SRF) (n=198) | 116

5. Secondary Outcome: Number of Patients With a Dry Retina (Neither IRF Nor SRF) up to Week 48 in the Study Eye
Description: Assessed by Spectral domain optical coherence tomography (SD-OCT) from the central reading center.
Time Frame: Baseline, Weeks 4, 8, 16, 48
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 289
Participants
  Baseline | 4
  Week 4 (n=260): number analyzed (Participants) | 260
  Week 4 (n=260) | 114
  Week 8 (n=229): number analyzed (Participants) | 229
  Week 8 (n=229) | 122
  Week 16 (n=222): number analyzed (Participants) | 222
  Week 16 (n=222) | 69
  Week 48 (n=198): number analyzed (Participants) | 198
  Week 48 (n=198) | 80

6. Secondary Outcome: Distribution of the Last Interval With no Disease Activity up to Week 48 in the Study Eye
Description: as for outcome 1
Time Frame: Intervals of 0,4,5,6,7,8,9,10,11,12,13,14,15,16,17 Weeks
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 289
Participants
  q0wk | 10
  q4wk | 24
  q5wk | 13
  q6wk | 7
  q7wk | 19
  q8wk | 102
  q9wk | 28
  q10wk | 10
  q11wk | 13
  q12wk | 29
  q13wk | 10
  q14wk | 3
  q15wk | 4
  q16wk | 13
  q17wk | 4

7. Secondary Outcome: Distribution of the Maximal Intervals With no Disease Activity up to Week 48 in the Study Eye
Description: as for outcome 1
Time Frame: Intervals of 0,4,5,6,7,8,9,10,11,12,13,14,15,16,17 Weeks
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 289
Participants
  q0wk | 10
  q4wk | 19
  q5wk | 18
  q6wk | 3
  q7wk | 6
  q8wk | 51
  q9wk | 48
  q10wk | 19
  q11wk | 14
  q12wk | 56
  q13wk | 16
  q14wk | 3
  q15wk | 5
  q16wk | 16
  q17wk | 4
  q20wk | 1

8. Secondary Outcome: Average Change in BCVA (Best-Corrected Visual Acuity) From Baseline up to Week 48 in the Study Eye
Description: BCVA was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  Visual Function of the study eye was assessed using the ETDRS protocol.
  Min and max possible scores are 0-100 respectively. A higher score represents better visual functioning.
Time Frame: Baseline, Weeks 4, 8, 16, 48
Population: Full Analysis Set - The full analysis set (FAS) comprises all patients who received at least one IVT injection of study treatment without protocol deviation with impact with at least one valid post baseline assessment.
Measure: Mean (Standard Deviation); unit: Letters read
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 259
Letters read
  Week 4 | 2.6 (6.09)
  Week 8 (n=231): number analyzed (Participants) | 231
  Week 8 (n=231) | 4.1 (6.68)
  Week 16 (n=218): number analyzed (Participants) | 218
  Week 16 (n=218) | 4.1 (7.41)
  Week 48 (n=199): number analyzed (Participants) | 199
  Week 48 (n=199) | 3.2 (9.22)

9. Secondary Outcome: Summary of Treatment-emergent Adverse Events - Overall
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study.
Time Frame: Adverse events were reported from first dose of study treatment until Week 48, plus 30 days post treatment, up to a maximum duration of 52 weeks.
Population: Safety Analysis Set (SAF) - Includes all patients who were randomized to treatment, which includes 6 patients who were randomized but not treated.
Measure: Count of Participants; unit: Participants
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 295
Participants
  Any adverse event | 165
  Any adverse event - Treatment-related | 34
  Any adverse event - Procedure-related | 33
  Serious adverse events | 28
  Serious adverse events- Treatment-related | 14
  Serious adverse events - Procedure-related | 4
  Fatal SAEs | 2
  Fatal SAEs - Treatment-related | 0
  Fatal SAEs - Procedure-related | 0
  AEs causing treatment discontinuation | 39
  AEs causing treatment discontinuation - Treatment-related | 30
  AEs causing treatment discontinuation - Procedure-related | 5
  AEs leading to treatment interruption | 0

10. Secondary Outcome: Summary of Treatment-emergent Adverse Events Regardless of Study Treatment Relationship by Primary System Organ Class, Preferred Term, and Maximum Severity - Ocular (Study Eye)
Description: as for outcome 9
Time Frame: as for outcome 9
Population: Safety Analysis Set (SAF) - Includes all patients who were randomized to treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 295
Participants
  Number of patients with at least one AE | 100
  Eye disorders | 92
  Eye disorders-Vitreous floaters | 15
  Eye disorders-Ocular hypertension | 11
  Eye disorders-Vitreous detachment | 9
  Eye disorders-Uveitis | 8
  Eye disorders-Vitritis | 8
  Eye disorders-Cataract | 5
  Eye disorders-Iridocyclitis | 5
  Eye disorders-Dry eye | 4
  Eye disorders-Eye inflammation | 4
  Eye disorders-Eye irritation | 4
  Eye disorders-Eye pain | 4
  Eye disorders-Posterior capsule opacification | 4
  Eye disorders-Retinal hemorrhage | 4
  Eye disorders-Vision blurred | 4
  Eye disorders-Conjunctival hemorrhage | 2
  Eye disorders-Ocular vasculitis | 2
  Eye disorders-Retinal artery occlusion | 2
  Eye disorders-Retinal occlusive vasculitis | 2
  Eye disorders-Retinal pigment epithelial tear | 2
  Eye disorders-Retinal tear | 2
  Eye disorders-Retinal vasculitis | 2
  Eye disorders-Visual acuity reduced | 2
  Eye disorders-Anterior chamber cell | 1
  Eye disorders-Cyclitis | 1
  Eye disorders-Diplopia | 1
  Eye disorders-Dyschromatopsia | 1
  Eye disorders-Eye hematoma | 1
  Eye disorders-Eye pruritus | 1
  Eye disorders-Glaucoma | 1
  Eye disorders-Keratitis | 1
  Eye disorders-Lacrimation increased | 1
  Eye disorders-Macular hole | 1
  Eye disorders-Ocular hyperemia | 1
  Eye disorders-Ocular ischemic syndrome | 1
  Eye disorders-Retinal aneurysm | 1
  Eye disorders-Retinal degeneration | 1
  Eye disorders-Retinal detachment | 1
  Eye disorders-Retinal drusen | 1
  Eye disorders-Retinal perivascular sheathing | 1
  Eye disorders-Serous retinal detachment | 1
  Eye disorders-Swelling of eyelid | 1
  Eye disorders-Visual field defect | 1
  Eye disorders-Vitreous hemorrhage | 1
  Eye disorders-Vitreous opacities | 1
  Infections and infestations | 3
  Infections and infestations-Conjunctivitis | 2
  Infections and infestations-Herpes ophthalmic | 1
  Injury, poisoning and procedural complications | 3
  Injury, poisoning and procedural complications-Foreign body in eye | 1
  Injury, poisoning and procedural complications-Procedural pain | 1
  Injury, poisoning and procedural complications-Thermal burn | 1
  Investigations | 7
  Investigations-Intraocular pressure increased | 7

11. Secondary Outcome: Summary of Treatment-emergent Adverse Events Regardless of Study Treatment Relationship by Primary System Organ Class, Preferred Term, and Maximum Severity - Non-ocular
Description: as for outcome 9
Time Frame: as for outcome 9
Population: Safety Analysis Set (SAF) - Includes all patients who were randomized to treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 295
Participants | 90

12. Post Hoc Outcome: All Collected Deaths
Description: On-treatment - up to 52 weeks; Post-treatment - greater than 30 days after last treatment, up to a maximum timeframe of 81 days after treatment
Time Frame: On-treatment - up to 52 weeks; Post-treatment - greater than 30 days after last treatment, up to 81 days post-treatment
Population: Safety Analysis Set (SAF) - Includes all patients who were randomized to treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 295
Participants
  On-Treatment Deaths | 0
  Post-Treatment Deaths | 2
  All Deaths | 2

ADVERSE EVENTS:
Time Frame: On treatment Adverse events are reported from first dose of study treatment until Week 48, plus 30 days post treatment, up to a maximum time period of 52 weeks. Post-treatment Adverse events are reported for the time period greater than 30 days after last treatment, up to 81 days post-treatment.
Description: Safety set
Arm/Group | RTH258/Brolucizumab
All-Cause Mortality (participants affected / at risk) | 2/295
Serious Adverse Events (participants affected / at risk) | 28/295
Other Adverse Events (participants affected / at risk) | 148/295
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RTH258/Brolucizumab (N=295)
Angina pectoris (Cardiac disorders) | 2
Cardiomyopathy (Cardiac disorders) | 1
Cyclitis - Study eye (Eye disorders) | 1
Eye haematoma - Study eye (Eye disorders) | 1
Eye inflammation - Study eye (Eye disorders) | 1
Iridocyclitis - Study eye (Eye disorders) | 1
Retinal artery occlusion - Study eye (Eye disorders) | 2
Retinal occlusive vasculitis - Study eye (Eye disorders) | 2
Uveitis - Study eye (Eye disorders) | 7
Vitritis - Study eye (Eye disorders) | 3
Chest pain (General disorders) | 1
Traumatic intracranial haematoma (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RTH258/Brolucizumab (N=295)
Arrhythmia (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Age-related macular degeneration - Fellow eye (Eye disorders) | 3
Anterior chamber cell - Study eye (Eye disorders) | 1
Blepharitis (Eye disorders) | 1
Cataract - Both eye (Eye disorders) | 4
Cataract - Fellow eye (Eye disorders) | 2
Cataract - Study eye (Eye disorders) | 1
Chalazion (Eye disorders) | 2
Conjunctival haemorrhage - Study eye (Eye disorders) | 2
Diplopia - Both eye (Eye disorders) | 1
Dry eye - Both eye (Eye disorders) | 1
Dry eye - Study eye (Eye disorders) | 1
Dyschromatopsia - Both eye (Eye disorders) | 1
Eye inflammation - Study eye (Eye disorders) | 3
Eye irritation - Both eye (Eye disorders) | 1
Eye irritation - Study eye (Eye disorders) | 3
Eye pain - Study eye (Eye disorders) | 3
Eye pruritus - Study eye (Eye disorders) | 1
Eyelid irritation (Eye disorders) | 1
Glaucoma - Both eye (Eye disorders) | 1
Iridocyclitis - Study eye (Eye disorders) | 4
Keratitis - Study eye (Eye disorders) | 1
Lacrimation increased - Both eye (Eye disorders) | 1
Macular hole - Study eye (Eye disorders) | 1
Neovascular age-related macular degeneration - Fellow eye (Eye disorders) | 11
Neovascular age-related macular degeneration - Study eye (Eye disorders) | 1
Ocular hyperaemia - Study eye (Eye disorders) | 1
Ocular hypertension - Both eye (Eye disorders) | 1
Ocular hypertension - Fellow eye (Eye disorders) | 1
Ocular hypertension - Study eye (Eye disorders) | 10
Ocular vasculitis - Study eye (Eye disorders) | 2
Posterior capsule opacification - Both eye (Eye disorders) | 1
Posterior capsule opacification - Fellow eye (Eye disorders) | 1
Posterior capsule opacification - Study eye (Eye disorders) | 3
Retinal degeneration - Study eye (Eye disorders) | 1
Retinal detachment - Study eye (Eye disorders) | 1
Retinal drusen - Study eye (Eye disorders) | 1
Retinal haemorrhage - Fellow eye (Eye disorders) | 1
Retinal haemorrhage - Study eye (Eye disorders) | 4
Retinal occlusive vasculitis - Study eye (Eye disorders) | 1
Retinal perivascular sheathing - Fellow eye (Eye disorders) | 1
Retinal perivascular sheathing - Study eye (Eye disorders) | 1
Retinal pigment epithelial tear - Study eye (Eye disorders) | 2
Retinal tear - Study eye (Eye disorders) | 2
Retinal vasculitis - Study eye (Eye disorders) | 2
Serous retinal detachment - Fellow eye (Eye disorders) | 1
Swelling of eyelid (Eye disorders) | 1
Uveitis - Study eye (Eye disorders) | 1
Vision blurred - Both eye (Eye disorders) | 1
Vision blurred - Fellow eye (Eye disorders) | 1
Vision blurred - Study eye (Eye disorders) | 3
Visual acuity reduced - Study eye (Eye disorders) | 2
Visual field defect - Study eye (Eye disorders) | 1
Vitreous detachment - Study eye (Eye disorders) | 9
Vitreous floaters - Both eye (Eye disorders) | 1
Vitreous floaters - Study eye (Eye disorders) | 12
Vitreous haemorrhage - Study eye (Eye disorders) | 1
Vitreous opacities - Study eye (Eye disorders) | 1
Vitritis - Study eye (Eye disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Gingival erosion (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Rectal polyp (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Allergy to arthropod sting (Immune system disorders) | 1
Allergy to synthetic fabric (Immune system disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Asymptomatic COVID-19 (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 4
COVID-19 (Infections and infestations) | 7
Conjunctivitis - Both eye (Infections and infestations) | 1
Conjunctivitis - Study eye (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Dermatophytosis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes ophthalmic - Study eye (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 3
Onychomycosis (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Periodontitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Foreign body in eye - Both eye (Injury, poisoning and procedural complications) | 1
Procedural pain - Study eye (Injury, poisoning and procedural complications) | 2
Spinal fracture (Injury, poisoning and procedural complications) | 1
Thermal burn - Both eye (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Intraocular pressure increased - Both eye (Investigations) | 1
Intraocular pressure increased - Study eye (Investigations) | 6
Prostatic specific antigen increased (Investigations) | 1
SARS-CoV-2 test positive (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Amnesia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Psychomotor skills impaired (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 1
Hallucination (Psychiatric disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal cyst (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract polyp (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Arterial stenosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 11
Hypotension (Vascular disorders) | 1
White coat hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT04264819/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/19/NCT04264819/SAP_001.pdf